CLINICAL TRIAL: NCT00890981
Title: A HR-pQCT Study in Postmenopausal Women Previously Treated With Denosumab
Brief Title: A High-resolution Peripheral Quantitative Computed Tomography Study in Postmenopausal Women Previously Treated With Denosumab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20080747
Record Dates: First submitted 2009-04-23; First posted 2009-04-30 (Estimated); Results first posted 2011-07-28 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Low Bone Mass; Low Bone Mineral Density; Osteoporosis; Postmenopausal Osteoporosis
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis; Osteoporosis, Postmenopausal | interventions — Absorptiometry, Photon; Denosumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other): Participants who were randomized to either denosumab or placebo in Study 20050179 and at least 12 months had elapsed from their 20050179 end-of-study visit had dual energy X-ray absorptiometry (DXA) of the forearm and HR-pQCT of the tibia and radius on Day 1 of this study. No study drug was administered.
  Interventions: Procedure: high-resolution peripheral quantitative computed tomography (HR-pQCT); Procedure: Dual energy X-ray absorptiometry (DXA); Biological: Denosumab; Drug: Placebo

INTERVENTIONS:
Procedure: high-resolution peripheral quantitative computed tomography (HR-pQCT) — Bone densitometry and microarchitecture assessments of the distal radius and the distal tibia by HR-pQCT on Day 1.
Procedure: Dual energy X-ray absorptiometry (DXA) — Bone densitometry assessments of the forearm by DXA on day 1.
Biological: Denosumab — Denosumab 60 mg subcutaneously every 6 months in the previous study
Drug: Placebo — Placebo to denosumab subcutaneously every 6 months in the previous study

SUMMARY:
To evaluate the combined effect of denosumab treatment and discontinuation on cortical thickness at the distal radius by High Resolution-Peripheral Quantitative Computed Tomography (HR-pQCT). Participants randomized to either denosumab or placebo in the 20050179 (NCT00293813) study who completed that study (ie, attended an end of study visit) can be included in this study. At least 12 months should have elapsed since the patient's 20050179 end of study visit.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory, postmenopausal women
* Randomized to either denosumab or placebo in the 20050179 (NCT00293813) study and completed that study (ie, attended an end of study visit)
* At least 12 months have elapsed since their end of 20050179 study visit
* Provide signed informed consent

Exclusion Criteria:

* Subjects who failed to receive both doses of denosumab (or SQ [subcutaneous] placebo) during the 20050179 study
* Subjects who were randomized to the alendronate arm during the 20050179 study
* Subjects diagnosed with any of the following conditions following completion of the 20050179 study:
* Hyperthyroidism
* Hyperparathyroidism
* Malignancy within the last 5 years (except cervical carcinoma in situ or basal cell carcinoma)
* Any condition that required chronic (greater than three months cumulative and greater than 5 mg/day) glucocorticoid therapy
* Other diseases which affect bone metabolism
* Self-reported alcohol or drug abuse within the previous 12 months
* Any disorder that, in the opinion of the investigator, may compromise the ability of the subject to give written informed consent and/or comply with study procedures
* Received any investigational product other than denosumab in two years before the screening visit.
* Received > 3 months (or equivalent) of osteoporosis treatment since having completed the 20050179 study.
* Current use of the following osteoporosis agents: bisphosphonates, calcitonin, fluoride, parathyroid hormone analogue, selective estrogen receptor modulators, systemic oral or transdermal estrogen (except vaginal preparations and estrogen creams which are acceptable), strontium or tibolone.
* Currently enrolled in or has not yet completed at least 1 month since ending other investigational device or drug trial(s) (other than Amgen trial 20080287), or subject is receiving other investigational agent(s).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2009-07; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] concept.747 Treatment/discontinuation on wrist.Journal-004521;
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject enrolled on 14-JUL-2009. The last subject enrolled on 12-MAY-2010
Groups:
- Previous Placebo Treatment Group: Participants who had previously received placebo and completed Study 20050179 (NCT00293813). No study drug was administered during this study.
- Previous Denosumab Treatment Group: Participants who had previously received denosumab and completed Study 20050179. No study drug was administered during this study.
Period: Overall Study
Arm/Group | Previous Placebo Treatment Group | Previous Denosumab Treatment Group
Started | 39 | 40
Completed | 39 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Previous Placebo Treatment Group: Participants who had previously received placebo and completed Study 20050179. No study drug was administered during this study.
- Total: Total of all reporting groups
Arm/Group | Previous Placebo Treatment Group | Previous Denosumab Treatment Group | Total
Number analyzed (Participants) | 39 | 40 | 79
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (5.8) | 63.4 (6.5) | 63.7 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 40 | 79
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants] | 39 | 40 | 79
Months since last dose in 20050179 [Mean (Standard Deviation); unit: Months] | 32.1 (2.5) | 32.2 (2.7) | 32.1 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From the Parent Study Baseline in Cortical Thickness at the Distal Radius by HR-pQCT
Description: Percent change from the 20050179 Baseline in cortical thickness at the distal radius as determined by high-resolution peripheral quantitative computed tomography (HR-pQCT) at an average of 32 months since the last subcutaneous dose of denosumab or placebo in study 20050179.
Time Frame: Baseline of Study 20050179 and Day 1 of this study. Study 20050179 duration was up to 12 months and the median time since completion of Study 20050179 was 32 months.
Population: Participants with observed data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Previous Placebo Treatment Group | Previous Denosumab Treatment Group
Number analyzed (Participants) | 39 | 37
Percent change | -5.5 [-8.3 to -2.8] | -1.8 [-4.8 to 1.2]
Statistical Analysis 1: Comparison: Previous Placebo Treatment Group vs Previous Denosumab Treatment Group; An analysis of covariance model was fit with main effects for randomized treatment in study 20050179, baseline value, time since last subcutaneous dose of denosumab or placebo in study 20050179 as a continuous variable, and the age stratification from 20050179. Model included linear, quadratic and cubic time terms with treatment-by-time interaction; Test type: Superiority or Other; p = 0.0766, ANCOVA; Mean Difference (Final Values) = 3.7, 95% CI [-0.4 to 7.8]

2. Secondary Outcome: Percent Change From the Parent Study Baseline in Total Bone Mineral Density (BMD) at the Distal Radius by HR-pQCT
Description: Percent change from the 20050179 Baseline in total BMD at the distal radius as determined by HR-pQCT at an average of 32 months since the last subcutaneous dose of denosumab or placebo in study 20050179.
Time Frame: as for outcome 1
Population: Participants with observed data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Previous Placebo Treatment Group | Previous Denosumab Treatment Group
Number analyzed (Participants) | 39 | 37
Percent change | -1.2 [-2.6 to 0.2] | 0.3 [-1.2 to 1.7]
Statistical Analysis 1: Comparison: Previous Placebo Treatment Group vs Previous Denosumab Treatment Group; An analysis of covariance model was fit with main effects for randomized treatment in study 20050179, baseline value, time since last subcutaneous dose of denosumab or placebo in study 20050179 as a continuous variable, and the age stratification from 20050179. Model included linear time term but without treatment-by-time interaction; Test type: Superiority or Other; p = 0.1648, ANCOVA; Mean Difference (Final Values) = 1.5, 95% CI [-0.6 to 3.5]

3. Secondary Outcome: Percent Change From the Parent Study Baseline in Cortical BMD at the Distal Radius by HR-pQCT
Description: Percent change from the 20050179 Baseline in cortical BMD at the distal radius as determined by HR-pQCT at an average of 32 months since the last subcutaneous dose of denosumab or placebo in study 20050179.
Time Frame: as for outcome 1
Population: Participants with observed data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Previous Placebo Treatment Group | Previous Denosumab Treatment Group
Number analyzed (Participants) | 39 | 37
Percent change | -1.0 [-1.7 to -0.3] | -0.0 [-0.8 to 0.8]
Statistical Analysis 1: Comparison: Previous Placebo Treatment Group vs Previous Denosumab Treatment Group; An analysis of covariance model was fit with main effects for randomized treatment in study 20050179, baseline value, time since last subcutaneous dose of denosumab or placebo in study 20050179 as a continuous variable, and the age stratification from 20050179. Model included linear, quadratic and cubic time terms but without treatment-by-time interaction; Test type: Superiority or Other; p = 0.0228, ANCOVA; Mean Difference (Final Values) = 0.9, 95% CI [0.1 to 1.7]

4. Secondary Outcome: Percent Change From the Parent Study Baseline in Trabecular BMD at the Distal Radius by HR-pQCT
Description: Percent change from the 20050179 Baseline in trabecular BMD at the distal radius as determined by HR-pQCT at an average of 32 months since last subcutaneous dose of denosumab or placebo in study 20050179.
Time Frame: as for outcome 1
Population: Participants with observed data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Previous Placebo Treatment Group | Previous Denosumab Treatment Group
Number analyzed (Participants) | 39 | 37
Percent change | 5.1 [2.3 to 8.0] | 5.9 [2.8 to 9.0]
Statistical Analysis 1: Comparison: Previous Placebo Treatment Group vs Previous Denosumab Treatment Group; An analysis of covariance model was fit with main effects for randomized treatment in study 20050179, baseline value, time since last subcutaneous dose of denosumab or placebo in study 20050179 as a continuous variable, and the age stratification from 20050179. Model includes linear, quadratic and cubic time terms but without treatment-by-time interaction; Test type: Superiority or Other; p = 0.6560, ANCOVA; Mean Difference (Final Values) = 0.7, 95% CI [-2.5 to 4.0]

5. Secondary Outcome: Percent Change From the Parent Study Baseline in Cortical Thickness at the Distal Tibia by HR-pQCT
Description: Percent change from the 20050179 Baseline in cortical thickness at the distal tibia as determined by HR-pQCT at an average of 32 months since the last subcutaneous dose of denosumab or placebo in study 20050179.
Time Frame: as for outcome 1
Population: Participants with observed data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Previous Placebo Treatment Group | Previous Denosumab Treatment Group
Number analyzed (Participants) | 39 | 40
Percent change | -6.4 [-7.8 to -5.1] | -4.6 [-5.9 to -3.3]
Statistical Analysis 1: Comparison: Previous Placebo Treatment Group vs Previous Denosumab Treatment Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0594, ANCOVA; Mean Difference (Final Values) = 1.8, 95% CI [-0.1 to 3.7]

6. Secondary Outcome: Percent Change From the Parent Study Baseline in Total BMD at the Distal Tibia by HR-pQCT
Description: Percent change from the 20050179 Baseline in total BMD at the distal tibia as determined by HR-pQCT at an average of 32 months since last subcutaneous dose of denosumab or placebo in study 20050179.
Time Frame: as for outcome 1
Population: Participants with observed data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Previous Placebo Treatment Group | Previous Denosumab Treatment Group
Number analyzed (Participants) | 39 | 40
Percent change | -1.6 [-2.8 to -0.4] | 1.0 [-0.2 to 2.2]
Statistical Analysis 1: Comparison: Previous Placebo Treatment Group vs Previous Denosumab Treatment Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0032, ANCOVA; Mean Difference (Final Values) = 2.6, 95% CI [0.9 to 4.3]

7. Secondary Outcome: Percent Change From the Parent Study Baseline in Cortical BMD at the Distal Tibia by HR-pQCT
Description: Percent change from the 20050179 Baseline in cortical BMD at the distal tibia as determined by HR-pQCT at an average of 32 months since the last subcutaneous dose of denosumab or placebo in study 20050179.
Time Frame: as for outcome 1
Population: Participants with observed data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Previous Placebo Treatment Group | Previous Denosumab Treatment Group
Number analyzed (Participants) | 39 | 40
Percent change | -1.0 [-1.7 to -0.3] | -0.6 [-1.4 to 0.2]
Statistical Analysis 1: Comparison: Previous Placebo Treatment Group vs Previous Denosumab Treatment Group; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.2897, ANCOVA; Mean Difference (Final Values) = 0.4, 95% CI [-0.4 to 1.2]

8. Secondary Outcome: Percent Change From the Parent Study Baseline in Trabecular BMD at the Distal Tibia by HR-pQCT
Description: Percent change from the 20050179 Baseline in trabecular BMD at the distal tibia as determined by HR-pQCT at an average of 32 months since the last subcutaneous dose of denosumab or placebo in study 20050179.
Time Frame: as for outcome 1
Population: Participants with observed data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Previous Placebo Treatment Group | Previous Denosumab Treatment Group
Number analyzed (Participants) | 39 | 40
Percent change | 2.9 [1.0 to 4.9] | 6.8 [4.9 to 8.8]
Statistical Analysis 1: Comparison: Previous Placebo Treatment Group vs Previous Denosumab Treatment Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0067, ANCOVA; Mean Difference (Final Values) = 3.9, 95% CI [1.1 to 6.7]

9. Secondary Outcome: Percent Change of Distal 1/3 Radius BMD From the Parent Study Baseline by DXA
Description: Percent change of distal 1/3 radius BMD from the 20050179 Baseline as determined by dual energy X-ray absorptiometry (DXA) at an average of 32 months since last subcutaneous dose of denosumab or placebo in study 20050179.
Time Frame: as for outcome 1
Population: Participants with observed data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Previous Placebo Treatment Group | Previous Denosumab Treatment Group
Number analyzed (Participants) | 39 | 40
Percent change | -2.0 [-3.3 to -0.8] | 0.0 [-1.2 to 1.2]
Statistical Analysis 1: Comparison: Previous Placebo Treatment Group vs Previous Denosumab Treatment Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0184, ANCOVA; Mean Difference (Final Values) = 2.1, 95% CI [0.4 to 3.8]

10. Secondary Outcome: Percent Change of Ultradistal Radius BMD From the Parent Study Baseline by DXA
Description: Percent change of ultradistal radius BMD from the 20050179 Baseline as determined by DXA at an average of 32 months since last the subcutaneous dose of denosumab or placebo in study 20050179.
Time Frame: as for outcome 1
Population: Participants with observed data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Previous Placebo Treatment Group | Previous Denosumab Treatment Group
Number analyzed (Participants) | 39 | 40
Percent change | -3.5 [-4.9 to -2.2] | -1.9 [-3.3 to -0.6]
Statistical Analysis 1: Comparison: Previous Placebo Treatment Group vs Previous Denosumab Treatment Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0911, ANCOVA; Mean Difference (Final Values) = 1.6, 95% CI [-0.3 to 3.5]

11. Secondary Outcome: Percent Change of Total Radius BMD From the Parent Study Baseline by DXA
Description: Percent change of total radius BMD from the 20050179 Baseline as determined by DXA at an average of 32 months since the last subcutaneous dose of denosumab or placebo in study 20050179.
Time Frame: as for outcome 1
Population: Participants with observed data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Previous Placebo Treatment Group | Previous Denosumab Treatment Group
Number analyzed (Participants) | 39 | 40
Percent change | -3.0 [-4.0 to -2.0] | -0.9 [-1.9 to 0.1]
Statistical Analysis 1: Comparison: Previous Placebo Treatment Group vs Previous Denosumab Treatment Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0035, ANCOVA; Mean Difference (Final Values) = 2.1, 95% CI [0.7 to 3.5]

12. Secondary Outcome: Actual Value of Serum Type I C-telopeptide
Description: Actual value of Serum Type I C-telopeptide measured from blood samples taken on Day 1 (an average of 32 months since the last subcutaneous dose of denosumab or placebo in study 20050179).
Time Frame: Day 1
Population: Participants with observed data.
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Previous Placebo Treatment Group | Previous Denosumab Treatment Group
Number analyzed (Participants) | 39 | 40
ng/mL | 0.6 [0.5 to 0.6] | 0.7 [0.6 to 0.7]
Statistical Analysis 1: Comparison: Previous Placebo Treatment Group vs Previous Denosumab Treatment Group; ANCOVA based on the log transformed actual values with main effects for randomized treatment in study 20050179, baseline value, time since last subcutaneous dose of denosumab or placebo in study 20050179 as a continuous variable, and the age stratification from 20050179. Model included linear time term but without treatment-by-time interaction; Test type: Superiority or Other; p = 0.0591, ANCOVA; Ratio of Denosumab to Placebo = 1.1, 95% CI [1.0 to 1.3]

13. Secondary Outcome: Actual Value of Procollagen Type 1 N-terminal Peptide
Description: Actual value of Type 1 N-terminal Peptide as measured from blood samples taken on Day 1 (an average of 32 months since the last subcutaneous dose of denosumab or placebo in study 20050179).
Time Frame: Day 1
Population: Participants with observed data.
Measure: Least Squares Mean (95% Confidence Interval); unit: µg/L
Arm/Group | Previous Placebo Treatment Group | Previous Denosumab Treatment Group
Number analyzed (Participants) | 39 | 40
µg/L | 49.8 [45.6 to 54.3] | 58.9 [54.1 to 64.2]
Statistical Analysis 1: Comparison: Previous Placebo Treatment Group vs Previous Denosumab Treatment Group; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.0079, ANCOVA; Ratio of Denosumab to Placebo = 1.2, 95% CI [1.0 to 1.3]

ADVERSE EVENTS:
Time Frame: AEs (serious only) were collected after informed consent and through 30 days after the study procedures, maximum time on study was 44 days.
Description: Only Serious Adverse Events were collected for this study.
Arm/Group | Previous Placebo Treatment Group | Previous Denosumab Treatment Group
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/40
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.